CLINICAL TRIAL: NCT03301324
Title: Intubation Assist Clinical Study
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 7701
Record Dates: First submitted 2017-09-21; First posted 2017-10-04 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Intubation, Intratracheal
Keywords: intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Intubation Assist Dashboard — The ZOLL X Series Intubation Assist Dashboard feature guides the operator through a three-step auscultation process to verify the proper placement of an endotracheal tube.

SUMMARY:
The Intubation Assist Clinical Study is an observational study of adult patients scheduled for elective surgery under general anesthesia to assess the user interface, assess transthoracic impedance by the ventilation volume and assess transthoracic impedance. Monitoring will begin at the time the patient is pre-oxygenated in preparation for endotracheal intubation and will continue until 30 minutes after intubation is achieved.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Requiring intubation and assisted ventilation
* Patient undergoing elective surgery
* Able to give informed consent

Exclusion Criteria:

* Skin condition that would interfere with electrodes
* Inability/failure to intubate
* Pregnancy
* Surgery that prevents the application of electrodes and monitoring equipment.
* Previous excision of complete or partial lung; congenital lung abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective surgery using general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Assessment of the user interface | Assessment will be made after using Intubation Assist approximately 30 minutes after successful intubation

SECONDARY OUTCOMES:
Assessment of transthoracic impedance | Impedance measurements will be collected during intubation and will not exceed 30 minutes from the start of intubation

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wik, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kramer-Johansen J, Eilevstjonn J, Olasveengen TM, Tomlinson AE, Dorph E, Steen PA. Transthoracic impedance changes as a tool to detect malpositioned tracheal tubes. Resuscitation. 2008 Jan;76(1):11-6. doi: 10.1016/j.resuscitation.2007.07.021. Epub 2007 Aug 23. PMID 17719166
- [Background] Losert H, Risdal M, Sterz F, Nysaether J, Kohler K, Eftestol T, Wandaller C, Myklebust H, Uray T, Sodeck G, Laggner AN. Thoracic impedance changes measured via defibrillator pads can monitor ventilation in critically ill patients and during cardiopulmonary resuscitation. Crit Care Med. 2006 Sep;34(9):2399-405. doi: 10.1097/01.CCM.0000235666.40378.60. PMID 16850000
- [Background] Roberts K, Srinivasan V, Niles DE, Eilevstjonn J, Tyler L, Boyle L, Bishnoi R, Ferry S, Nysaether J, Stavland M, Litman RS, Helfaer M, Nadkarni V. Does change in thoracic impedance measured via defibrillator electrode pads accurately detect ventilation breaths in children? Resuscitation. 2010 Nov;81(11):1544-9. doi: 10.1016/j.resuscitation.2010.07.010. Epub 2010 Aug 25. PMID 20800333
- [Background] Hamilton LH, Beard JD, Kory RC. Impedance measurement of tidal volume and ventilation. J Appl Physiol. 1965 May;20(3):565-8. doi: 10.1152/jappl.1965.20.3.565. No abstract available. PMID 5837579
- [Background] Mort TC. Emergency tracheal intubation: complications associated with repeated laryngoscopic attempts. Anesth Analg. 2004 Aug;99(2):607-13, table of contents. doi: 10.1213/01.ANE.0000122825.04923.15. PMID 15271750
- [Background] Jaber S, Amraoui J, Lefrant JY, Arich C, Cohendy R, Landreau L, Calvet Y, Capdevila X, Mahamat A, Eledjam JJ. Clinical practice and risk factors for immediate complications of endotracheal intubation in the intensive care unit: a prospective, multiple-center study. Crit Care Med. 2006 Sep;34(9):2355-61. doi: 10.1097/01.CCM.0000233879.58720.87. PMID 16850003